CLINICAL TRIAL: NCT00247078
Title: The Efficacy and Safety of Aracmyn® [Antivenin Latrodectus (Black Widow)Equine Immune F(ab)2], in Patients With Systemic Latrodectism: A Phase II, Multi-center, Randomized, Double-Blind Trial
Brief Title: The Efficacy and Safety of Aracmyn in Patients With Systemic Latrodectism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Bioclon S.A. de C.V. (Industry)
Collaborators: Rocky Mountain Poison and Drug Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR-03/02
Record Dates: First submitted 2005-10-28; First posted 2005-11-01 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Arachnidism; Latrodectism
Keywords: black; widow; spider; antivenom
MeSH Terms: conditions — Spider Bites

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients with moderate or severe pain due to Black Widow envenomation
  Interventions: Biological: widow spider antivenom
- 2 (Placebo Comparator): Patients with moderate to severe pain due to Black Widow envenomation
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: widow spider antivenom — 3 vials of antivenom capable of neutralizing 600 LD50 of L. mactans
  Other Names: Analatro
  Arms: 1
Biological: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of an investigational antivenom and the current standard of care (pain management with opioid analgesics) for treating patients with a widow spider bite. The working hypotheses are as follows:

1. the investigational antivenom is more promptly effective at alleviating the pain associated with a widow spider bite than routine management with opioid pain medication
2. the investigational antivenom is as safe a treatment as opioid pain medication in treating patients with a widow spider bite.

DETAILED DESCRIPTION:
The purpose of this randomized, double-blind, multi-center phase II trial is to examine the safety and efficacy of Aracmyn® [Antivenin Latrodectus (Black Widow) Equine Immune F(ab)2], a new antivenom, for treatment of patients envenomed by the widow spider. Twenty-four subjects will be randomized to receive either the study drug or control (normal saline) through intravenous (IV) infusion. Following infusion, subjects will be monitored for changes in pain and clinical signs during a two-hour observation period. A standard dose of IV fentanyl will be offered to all subjects as pain medication at specific intervals following treatment. Vital signs, blood samples, and pain intensity scores (using a visual analog scale, VAS) will be collected before and after the infusion, as well as during the observation period. This study uses a treatment failure protocol, which involves administration of Merck Antivenin to subjects who do not obtain adequate pain relief from the study drug or control. Primary efficacy and safety endpoints for this 12-month trial will be improvement in pain intensity and clinical signs and incidence of adverse events, respectively.

ELIGIBILITY:
Inclusion Criteria:

* patient presents for treatment within 72 hours from time of symptoms onset
* clinical diagnosis of widow spider envenomation
* patient has moderate to severe pain intensity

Exclusion Criteria:

* history of significant cardiac, respiratory, hepatic, or renal disease
* distracting injury or chronic pain syndrome that would obscure pain intensity assessment
* history of asthma or known sensitivity to fentanyl, morphine, diazepam, or equine serum
* pregnant or lactating

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-10; Primary Completion 2006-10 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
between-treatment groups difference in pain intensity (pre- and post-treatment) | within first two hours

SECONDARY OUTCOMES:
between-treatment groups difference in proportion of treatment failures (absence of pain relief or return to hospital) | within 24 hours after discharge from emergency department
between-treatment groups difference in incidence of drug-related adverse events. | onset of adverse events within 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Dart, MD PhD, Principal Investigator — Rocky Mountain Poison and Drug Center; Walter Garcia, MD, Study Director — Instituto Bioclon S.A. de C.V.
Locations (1):
- Denver Health and Hospital Authority, Denver, Colorado, United States